CLINICAL TRIAL: NCT04048434
Title: Effectivity of Extracorporeal Cytokine Adsorption (Cytosorb) as Additive Treatment of CAR-T Cell Associated Cytokine Release (CRS) Syndrome and Encephalopathy Syndrome (CRES)
Brief Title: Extracorporeal Cytokine Adsorption as Additive Treatment of CAR-T Associated Cytokine Release Syndrome (CRS)
Acronym: CYTORELEASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRS01
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cytokine Release Syndrome; CAR-T
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care (SOC) (No Intervention)
- Cyotosorb (Experimental)
  Interventions: Device: Cytosorb

INTERVENTIONS:
Device: Cytosorb — extracorporeal cytokine adsorption
  Arms: Cyotosorb

SUMMARY:
Patients with severe CAR-T cell associated cytokine release syndrome (CRS) (defined as vasopressor dependent) will be treated with standard of care (SOC) + cytokine adsorption (6hourly for 24 hrs).

Primary endpoint is the change in plasma IL-6 between 0 and 24 hrs.

ELIGIBILITY:
Inclusion Criteria:

* severe CRS (> 3) and / or severe CRES (>3)

AND

- CRS/CRES onset < 6 hrs

Exclusion Criteria:

* Heparine allergy
* contraindication for anticoagulation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
IL-6 change | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sascha David, MD, Principal Investigator — Hannover Medical School
Locations (2):
- Hannover Medical School, Hanover, Germany
- Universitätsspital Zürich (USZ), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stahl K, Schmidt BMW, Hoeper MM, Skripuletz T, Mohn N, Beutel G, Eder M, Welte T, Ganser A, Falk CS, Koenecke C, David S. Extracorporeal cytokine removal in severe CAR-T cell associated cytokine release syndrome. J Crit Care. 2020 Jun;57:124-129. doi: 10.1016/j.jcrc.2020.02.010. Epub 2020 Feb 19. PMID 32113143